CLINICAL TRIAL: NCT00082368
Title: A Pilot Study of Tc-94m Sestamibi PET MDR Imaging
Brief Title: PET Imaging With Tc-94m Sestamibi to Assess Resistance to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Choyke, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 040177; 04-C-0177; NCT00086853 (obsolete NCT alias)
Record Dates: First submitted 2006-07-07; First posted 2004-05-06 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Cancer
Keywords: Tariquidar; PET; Sestamibi; Cancer
MeSH Terms: conditions — Neoplasms | interventions — tariquidar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET (positron emission imaging) Imaging with Tc-94m Sestamibi (Experimental): PET sestamibi scans followed by tariquidar and repeat imaging
  Interventions: Drug: Tariquidar; Drug: Tc-94m Sestamibi

INTERVENTIONS:
Drug: Tariquidar — 3 days after initial PET patients will receive tariquidar and repeat imaging.
Drug: Tc-94m Sestamibi — Patients over 18 years of age, who are eligible for, or have completed enrollment in an active NCI (National Cancer Institute) protocol for treatment of cancer will undergo a PET sestamibi scan

SUMMARY:
Background:

* Tc-94m sestamibi is a radioactive imaging drug approved by the Food and Drug Administration to help photograph and study bodily functions.
* Tc-94m sestamibi accumulates in tumor cells and is eliminated from them in much the same way that some chemotherapy drugs are eliminated from cancer cells in patients with drug resistance.
* P-glycoprotein is a protein found on the surface of some cancer cells. The protein causes the cells to pump out, or reject, some types of chemotherapy drugs. P-glycoprotein also makes the cells reject sestamibi.
* Some drugs, including a drug called tariquidar, may block the pumping action of P-glycoprotein, giving the chemotherapy more time to work. Tariquidar can also help sestamibi stay in the cells longer.

Objectives:

-To evaluate the use of sestamibi for determining if chemotherapy is being rejected and if enough of the blocking drugs are present to stop the rejection.

Eligibility:

-Patients18 years of age and older with a tumor 2 cm or larger who are enrolled in or are eligible for enrollment in an active National Cancer Institute treatment protocol.

Design:

* Patients have two scans, one before receiving any drugs and a second 1-2 hours after receiving tariquidar. The second scan is done 72 or more hours after the first. For both scans, Tc-94m sestamibi is injected into a vein and a series of pictures are taken with an imaging camera called a PET (positron emission tomography) scanner. The pictures show where the sestamibi distributes in the body and monitors the effects of tariquidar on drug resistance. Blood samples are collected during the scan to examine the effect of tariquidar on P-glycoprotein in normal cells.
* Some patients may be asked to undergo a tumor biopsy to test for the presence of the P-glycoprotein on their cancer cells. This will be requested only in patients whose tumor is easily accessible and in whom a biopsy can be done with minimal risk.

DETAILED DESCRIPTION:
Background:

* A pilot study of PET imaging with Tc-94m sestamibi to assess activity of the multidrug transporter, MDR-1 (Multi Drug Resistance Protein 1)/P-glycoprotein, an ATP (adenosine 5'-triphosphate)-binding cassette protein that transports drug out of the cell, thereby reducing intracellular drug accumulation.
* Tariquidar is a safe, nontoxic antagonist of P-glycoprotein. Previous studies demonstrated that tariquidar increased retention of the radioimaging agent, Tc99 sestamibi in normal liver and in a subset of tumors. These studies were limited by the semiquantitative nature of total body imaging by conventional radionuclide scintigraphy
* In collaboration with the Clinical Center Nuclear Medicine Department, a PET imaging agent has been developed, Tc-94m sestamibi, and the FDA (Food and Drug Administration) has granted approval for its use in humans.

Objectives:

-To evaluate the feasibility of Tc-94m sestamibi as a PET imaging agent, which should allow greater resolution and quantitation and thereby make possible direct quantitative comparisons of tumor uptake before and after treatment with a P-glycoprotein antagonist.

Eligibility:

* Patients over 18 years of age, who are eligible for, or have completed enrollment in an active NCI (National Cancer Institute) protocol for treatment of cancer.
* Negative pregnancy test within 24 hrs of Tc-94m injection.
* An index lesion greater than 2cm will be required to optimize the PET images.
* Prior treatment with a P-glycoprotein antagonist is allowed.

Design:

* Designed as a feasibility study. Patients meeting the eligibility criteria and signing informed consent will undergo a PET sestamibi imaging scan in the Department of Nuclear Medicine. Seventy-two hours later, a dose of tariquidar will be administered before a repeat imaging study.
* Blood will be obtained for analysis of the pharmacokinetics of Tc-94m sestamibi, and for isolation of peripheral blood mononuclear cells to assay P-glycoprotein inhibition in circulating CD56+ cells. These assessments are needed to confirm the impact of tariquidar on P-glycoprotein in normal cells - for example, those involved in drug excretion and in circulating mononuclear cells. These results will then be used to inform the findings in the PET imaging study.
* Fifteen patients will be enrolled and pairwise comparisons will be made between the sestamibi residence times in tumor, normal liver, kidney, and heart. All comparisons are noted to be exploratory.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must be eligible for enrollment in an active NCI (National Cancer Institute) protocol for treatment of cancer.

Patients greater than or equal to 18 years old.

Performance Status ECOG (Eastern Cooperative Oncology Group) 0 - 2.

Patients must be able to give informed consent.

Women of childbearing potential must have a negative pregnancy test within 24 hrs of Tc-94m injection.

Patients who have previously received tariquidar will be eligible, since no study has systematically shown loss of MDR-1 (Multi Drug Resistance Protein 1)/Pgp expression in tumors following exposure to both tariquidar and an anticancer agent.

An index lesion greater than 1.5 cm will be required to optimize the PET (positron emission imaging) images.

EXCLUSION CRITERIA:

Patients who are pregnant or breast-feeding will not be enrolled in order to prevent radiation exposure in the developing fetus or infant.

Patients weighing greater than 136 kg (the weight limit for the scanner table).

Patients having only tumor sizes less than 1.5 cm will be excluded.

HIV (human immunodeficiency virus) positive patients will be excluded to prevent potential drug interactions between tariquidar and antiretroviral agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-05-16 (Actual); Primary Completion 2014-04-14 (Actual); Study Completion 2014-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Choyke, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Advani R, Saba HI, Tallman MS, Rowe JM, Wiernik PH, Ramek J, Dugan K, Lum B, Villena J, Davis E, Paietta E, Litchman M, Sikic BI, Greenberg PL. Treatment of refractory and relapsed acute myelogenous leukemia with combination chemotherapy plus the multidrug resistance modulator PSC 833 (Valspodar). Blood. 1999 Feb 1;93(3):787-95. PMID 9920827
- [Background] Agrawal M, Abraham J, Balis FM, Edgerly M, Stein WD, Bates S, Fojo T, Chen CC. Increased 99mTc-sestamibi accumulation in normal liver and drug-resistant tumors after the administration of the glycoprotein inhibitor, XR9576. Clin Cancer Res. 2003 Feb;9(2):650-6. PMID 12576431
- [Background] Bakker M, van der Graaf WT, Piers DA, Franssen EJ, Groen HJ, Smit EF, Kool W, Hollema H, Muller EA, De Vries EG. 99mTc-Sestamibi scanning with SDZ PSC 833 as a functional detection method for resistance modulation in patients with solid tumours. Anticancer Res. 1999 May-Jun;19(3B):2349-53. PMID 10472354
- [Background] Chen CC, Meadows B, Regis J, Kalafsky G, Fojo T, Carrasquillo JA, Bates SE. Detection of in vivo P-glycoprotein inhibition by PSC 833 using Tc-99m sestamibi. Clin Cancer Res. 1997 Apr;3(4):545-52. PMID 9815718
- [Background] Bates SE, Bakke S, Kang M, Robey RW, Zhai S, Thambi P, Chen CC, Patil S, Smith T, Steinberg SM, Merino M, Goldspiel B, Meadows B, Stein WD, Choyke P, Balis F, Figg WD, Fojo T. A phase I/II study of infusional vinblastine with the P-glycoprotein antagonist valspodar (PSC 833) in renal cell carcinoma. Clin Cancer Res. 2004 Jul 15;10(14):4724-33. doi: 10.1158/1078-0432.CCR-0829-03. PMID 15269145
- [Background] Kelly RJ, Robey RW, Chen CC, Draper D, Luchenko V, Barnett D, Oldham RK, Caluag Z, Frye AR, Steinberg SM, Fojo T, Bates SE. A pharmacodynamic study of the P-glycoprotein antagonist CBT-1(R) in combination with paclitaxel in solid tumors. Oncologist. 2012;17(4):512. doi: 10.1634/theoncologist.2012-0080. Epub 2012 Mar 13. PMID 22416063
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-C-0177.html

RESULTS

PARTICIPANT FLOW:
Groups:
- PET Imaging With Tc-94m Sestamibi: Positron Emission Tomography (PET) sestamibi scans followed by tariquidar and repeat imaging
  Tariquidar: 3 days after initial PET patients will receive tariquidar and repeat imaging.
  Tc-94m Sestamibi: Patients over 18 years of age, who are eligible for, or have completed enrollment in an active National Cancer Institute (NCI) protocol for treatment of cancer will undergo a PET sestamibi scan
Period: Overall Study
Arm/Group | PET Imaging With Tc-94m Sestamibi
Started | 12
Completed | 11
Not Completed | 1
Not completed — Not treated-pt had poor IV access | 1

BASELINE CHARACTERISTICS:
Arm/Group | PET Imaging With Tc-94m Sestamibi
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.82 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Performance Status: Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG Performance Status: Grade 0 is normal activity. Fully active, able to carry on all pre-disease performance without restriction. Grade 1 is symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). Grade 2 is in bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Grade 3 is in bed >50% of the time. Capable of only limited self-care. Grade 4 is 100% bedridden. Completely disabled. Grade 5 is dead.
  Participants
    Performance status: 0 | 2
    Performance status: 1 | 9
    Performance status: 2 | 1
    Performance status: 3 | 0
Histology [Count of Participants; unit: Participants]
  Colorectal cancer | 4
  Pancreatic cancer | 2
  Small cell lung cancer | 2
  Non-small cell lung cancer | 1
  Esophageal cancer | 1
  Prostate cancer | 1
  Ovarian cancer | 1
Prior Chemotherapy [Mean (Full Range); unit: prior therapies] | 3.5 [1 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Tc-94m Sestamibi Body Weight Standardized Uptake Value (SUV) Maximum in Tumor Tissue Before and After Administration of Tariquidar, a P-glycoprotein Antagonist.
Description: Sestamibi is a Pgp substrate that may be a surrogate for measuring drug efflux from tumors. Significant increase in the SUV in tumor is +25% over baseline.
Time Frame: 3 days
Measure: Mean (Full Range); unit: % change in Tc-94m Sestamibi SUVmax
Arm/Group | PET Imaging With Tc-94m Sestamibi
Number analyzed (Participants) | 12
% change in Tc-94m Sestamibi SUVmax | 44 [-10 to 153]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 69 months
Measure: Number; unit: participants
Arm/Group | PET Imaging With Tc-94m Sestamibi
Number analyzed (Participants) | 12
participants | 8

ADVERSE EVENTS:
Time Frame: 69 months
Arm/Group | PET Imaging With Tc-94m Sestamibi
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET Imaging With Tc-94m Sestamibi (N=12)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (5)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (2)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 1 (2)
Low Hemoglobin (Blood and lymphatic system disorders) | 4 (5)
Low Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (4)
Pain::Head/headache (Nervous system disorders) | 1 (1)
Low Platelets (Blood and lymphatic system disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The lack of flexibility around patient chemotherapy schedules made the protocol difficult to conduct. Future studies should make imaging integral to the treatment protocol .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No